CLINICAL TRIAL: NCT05394194
Title: Dosimetric Comparison of Three Radiation Techniques for Hypofractionated Whole Breast Radiotherapy in Early Breast Cancer
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Alshaymaa Abdelghaffar, Lecturer of Clinical Oncology, Sohag University
Other Study IDs: Soh-Med-22-05-24
Record Dates: First submitted 2022-05-24; First posted 2022-05-27 (Actual); Last update posted 2022-05-27 (Actual); Status verified 2022-05

CONDITIONS: Breast Cancer
Keywords: computer assisted, radiotherapy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- 3DCRT group: In this plan, we will create plans using three dimensional conformal radiotherapy, evaluate organs at risk doses, dose homogeneity and planned target volume coverage. Then compare these parameters with the two other plans.
- IMRT group: In this plan, we will create plans using intensity modulated radiotherapy (IMRT), evaluate organs at risk doses, dose homogeneity and planned target volume coverage. Then compare these parameters with the two other plans.
- VMAT plan: In this plan, we will create plans using volumetric modulated radiotherapy (VMAT), evaluate organs at risk doses, dose homogeneity and planned target volume coverage. Then compare these parameters with the two other plans.

SUMMARY:
We aim to compare three different radiation delivery techniques, namely three-dimensional conformal radiation therapy (3D-CRT), intensity modulated radiotherapy (IMRT) and volumetric modulated radiation therapy (VMAT) in left-sided early breast cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* left sided early breast cancer patients. Should have histopathological prove to have invasive breast cancer. Operated by breast conservative surgery. Have no associated comorbidities

Exclusion Criteria:

* locally advanced breast cancer. Patients who have total mastectomy. Patients who had previous chest irradiation or known comorbidities.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: 30 Female patients who will present to clinical Oncology department with early breast cancer, with pathological staging ≤ T2N0M0 and are operated by conservative breast surgery will be included in our current study.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2022-07-20 (Estimated); Primary Completion 2024-07-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Comparison of coverage of planned target volume(PTV) among the three plans. | 1 year
  PTV coverage in dose is compared among the three plans.
Comparison of doses to organs at risk among the three plans. | 1 year
  mean dose of the heart, lung volume receiving 20Gy, esophageal doses will be compared among the three plans

SECONDARY OUTCOMES:
Comparison of target homogeneity among the three plans. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Alshaymaa Abdelghaffar, PhD, Principal Investigator — Sohag University